CLINICAL TRIAL: NCT04182178
Title: Long-term Follow-up of Patient Satisfaction, Reflux Control and Gastrointestinal Disorders in Patients Undergoing Laparoscopic Surgical Treatment for GERD, With Partial or Total Fundoplication
Brief Title: Long-term Follow-up After Surgical Treatment for GERD (Gastroesophageal Reflux Disease)
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anders Thorell, Professor, Karolinska Institutet
Other Study IDs: 2019-03655
Record Dates: First submitted 2019-11-07; First posted 2019-12-02 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Patient Satisfaction; Relapse; Dysphagia; Bloating
MeSH Terms: conditions — Patient Satisfaction; Recurrence; Deglutition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gastroesophageal reflux: Laparoscopic total (Nissen) or posterior 270 degree (Toupét) partial fundoplication for the treatment of gastroesophageal reflux disease.
  Interventions: Other: 10 years follow up

INTERVENTIONS:
Other: 10 years follow up — Questionnaires

SUMMARY:
10 years of follow-up with SF-36 global (Quality of Life issues), GSRS (Gastrointestinal Symptom Rating Scale) and two reflux specific questionnaires.

DETAILED DESCRIPTION:
Long-term follow up with questionnaires after surgery with laparoscopic 270 degrees posterial partial fundoplication vs total fundoplication for the treatment of gastroesophageal reflux disease.

Quality of Life SF-36; physical and mental component scores. GSRS, five dimensions of abdominal symptoms; reflux, abdominal pain, indigestion, obstipation and diarrhea.

Reflux specificquestionnaries on various issues of reflux disease and frequency issues about reflux disease problems.

ELIGIBILITY:
Inclusion Criteria:

Gastroesophageal Reflux 10 years follow-up after surgery informed consent

Exclusion Criteria:

Deceased patients patients who declined participation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastroesophageal Reflux Disease
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
SF-36 Quality of life | 10 years
  The SF-36 It is comprised of 36 items that assess eight health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions. Physical and mental health summary scores are also derived from the eight RAND-36 scales. Higher scores mean a better outcome.
Gastrointestinal Symptom Rating Scale (GSRS) | 10 years after operation
  GSRS Gastrointestinal Symptom Rating Scale Scoring;The questionnaire, which contains 15 items, uses a seven-graded Likert scale, where 1 represents the most positive option and 7 the most negative one.
  A mean value for the items in each dimension should be calculated:
  Diarrhoea syndrome: 11. Increased passage of stools 12. Loose stools 14. Urgent need for defecation Indigestion syndrome: 6. Borborygmus 7. Abdominal distension 8. Eructation 9. Increased flatus Constipation syndrome: 10. Decreased passage of stools 13. Hard stools 15. Feeling of incomplete evacuation.
  Abdominal pain syndrome: 1. Abdominal pain 4. Sucking sensations 5. Nausea and vomiting Reflux syndrome: 2. Heartburn 3. Acid regurgitation

CONTACTS AND LOCATIONS:
Overall Officials: Anders Thorell, professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Ersta Hospital, Stockholm, Region Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Analatos A, Hakanson BS, Ansorge C, Lindblad M, Lundell L, Thorell A. Clinical Outcomes of a Laparoscopic Total vs a 270 degrees Posterior Partial Fundoplication in Chronic Gastroesophageal Reflux Disease: A Randomized Clinical Trial. JAMA Surg. 2022 Jun 1;157(6):473-480. doi: 10.1001/jamasurg.2022.0805. PMID 35442430